CLINICAL TRIAL: NCT05498636
Title: Selinexor Combined With Prednisone, Etoposide, and Lenalidomide as Introductive Treatment Following Immune-chemotherapy as Consolidated Therapy for Refractory Diffuse Large B-cell Lymphoma With p53 and/or c-Myc Expression
Brief Title: SPEL as Introductive Treatment Following Immune-chemotherapy as Consolidated Therapy for R/R DLBCL With p53 and/or c-Myc Expression
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202201
Record Dates: First submitted 2022-08-03; First posted 2022-08-12 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: DLBCL
Keywords: DLBCL; p53; c-myc; selinexor; lenalidomide; refractory/relapse
MeSH Terms: conditions — Recurrence | interventions — Prednisone; Etoposide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SPEL (Experimental)
  Interventions: Combination Product: Selinexor combined with Prednisone, Etoposide, and Lenalidomide

INTERVENTIONS:
Combination Product: Selinexor combined with Prednisone, Etoposide, and Lenalidomide — Selinexor combined with Prednisone, Etoposide, and Lenalidomide

SUMMARY:
This study is a phase II multi-center prospective clinical trail which investigates the efficacy and safety of Selinexor combined with prednisone, etoposide and lenalidomide in the treatment of relapsed/refractory diffuse large B-cell lymphoma (DLBCL) patient with high p53 and/or c-myc expression.

ELIGIBILITY:
Inclusion Criteria:

1. Any of the following as defined by the WHO, 2016 lymphoid neoplasm classifications and histologically confirmed：Diffuse large B-cell lymphoma with p53 and/ or c-Myc protein overexpression.

   Note: a. The cutoff value for p53 protein overexpression by immunohistochemistry (IHC) is 50%; cutoff value for c-Myc protein overexpression is 30-40%; b. For patients with high expression of C-Myc, dual-color FISH probes detection method should be used to check whether there is Myc and BCL2 gene rearrangement, which is cut by 5%; c. We need 5-10 pathological white films with a thickness of 5-10 um for review.
2. Patients who cannot tolerate or are unwilling to undergo intensive salvage therapy due to age or frailty; patients who have received at most three prior lines of regimen, in which stem cell transplantation is considered first-line.
3. With a life expectancy of ≥ 3 months
4. Age ≥ 18 years
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
6. At least 1 evaluable or measurable lesion that meets Lugano2014 criteria [Evaluable lesions: PET/CT examination showed increased uptake in lymph nodes or extranodal areas (higher than that in the liver), and pet/ct features were consistent with lymphoma. Measurable disease: Nodular lesions with longest diameter (LDi) greater than > 15mm or extranodal lesion with LDi >10mm. and FDG-PET positive lesions]
7. All screening laboratory tests should be performed according to the protocol and within 14 days before enrollment. Screening laboratory values must meet the following criteria： Routine blood tests (no blood transfusion, no G-CSF, no drug correction within 14 days before screening) : a. Hb≥80g/L；b.ANC≥1.0×109/L；c.PLT≥75×109/L.

   Blood biochemistry: a.TBIL≤1.5×upper limit of normal (ULN), or TBIL≤3×ULN(if due to liver involvement); b. ALT and AST≤3×ULN, or AST and ALT≤5.0 x ULN(if due to liver involvement); c. Serum creatinine ≤1.5×ULN, or Estimated creatinine clearance ≥ 50 mL/min (calculated using the formula of Cockcroft-Gault).

   Coagulation function (unless the subject is receiving anticoagulant treatment and the coagulation parameters (PT/INR and APTT) are within the expected range of anticoagulant treatment at the time of screening): INR≤1.5×ULN; APTT≤1.5×ULN.
8. Written informed consent of the patient

Exclusion Criteria:

1. Patient with hemophagocytic syndrome
2. With uncontrolled serious active infections, including active tuberculosis
3. Known to have central nervous system (CNS), testicular, breast lymphoma; Patients with massive pleural and peritoneal effusion
4. Previous treatment with Selinexor or lenalidomide in the past 6 months
5. Previous treatment with allogeneic hematopoietic stem cell transplantation or allogeneic organ transplantation.
6. Autologous hematopoietic stem cell transplantation was performed within 6 months prior to initiation of treatment.
7. Major surgery <28 days of C1D1.
8. Live vaccine (excluding attenuated influenza vaccine) within 28 days before study treatment.
9. Ongoing participation in another clinical study, or planned initiation of treatment in this study less than 4 weeks from the end of treatment in the previous clinical study.
10. Patients with serious medical diseases, such as organic heart disease, resulting in clinical symptoms or cardiac dysfunction (≥NYHA grade 2), a history of myocardial infarction within 6 months prior to screening, echocardiographic ejection fraction < 50%, and severe thromboembolic diseases.
11. Positive HIV serologies before inclusion.
12. Other malignant tumors in the past 5 years, except basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, and gastrointestinal intramucosal carcinoma after radical treatment.
13. Additional systemic antitumor therapy may be accepted during the study period.
14. Other conditions that patients considered unsuitable for inclusion by the researchers.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
CR rate | At the end of Cycle 4 (each cycle is 28 days)
  complete remission rate after 4 cycles of SPEL regimen
ORR | At the end of Cycle 4 (each cycle is 28 days)
  overall response rate after 4 cycles of SPEL regimen

SECONDARY OUTCOMES:
AE | from the first dose of SPEL regimen to 3 months after last dose of the regimen
  adverse event of SPEL regimen

CONTACTS AND LOCATIONS:
Locations (1):
- the affiliated hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No